CLINICAL TRIAL: NCT02975986
Title: Renal Uptake of Fatty Acids (FFA) in Patients With Idiopathic Uric Acid Nephrolithiasis (IUAN)
Acronym: IUAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 092014-032; R01DK081423-07 (NIH)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Uric Acid Nephrolithiasis
Keywords: Nephrolithiasis, Uric Acid; Fatty Acid
MeSH Terms: conditions — Nephrolithiasis | interventions — Technetium Tc 99m Mertiatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled metabolic diet (Other): All study patients will be placed on an instructed controlled metabolic diet. Intervention: Uptake of radioactive isotope by the kidney Radiotracer: 123I-BMIPP, 99mTc-MAG3
  Interventions: Other: 123I-BMIPP; Other: 99mTc-MAG3

INTERVENTIONS:
Other: 123I-BMIPP — Uptake of radioactive isotope by the kidney
Other: 99mTc-MAG3 — Uptake of radioactive isotope by the kidney

SUMMARY:
The investigators will test the hypothesis that renal uptake of free (i.e. non-esterified) fatty acids (FFa) is increased in iuan. To accomplish this goal the investigators will measure renal FFa uptake FFa uptake in vivo in patients with iuan and matched non-stone forming subjects via single-photon emission computed tomography (SPeCT)/CT imaging.

The definitive proof of the hypothesis rests on whether increased renal FFa uptake is demonstrable in humans with iuan.

DETAILED DESCRIPTION:
This is a cross-sectional study of patients with iuan and matched non-stone formers to test the hypothesis that renal FFa uptake is increased in iuan, using noninvasive 123i-labeled [MiCRo-SYMBoL]-methyl-p-iodo-phenyl-pentadecanoic acid(123i-BMiPP) SPeCT/CT imaging, an established FFa analog approved for human studies.

Participants will be placed on an instructed controlled metabolic diet (30% fat, 15% protein, 55% carbohydrate, 300 mg cholesterol per day, 400 mg calcium, 800mg phosphorus, 100 meq sodium, with low acid ash content, and 3000 cc distilled water) for 5 days to exclude dietary confounders (3 days as outpatient and the final 2 days as inpatient). On days 4 and 5, two fasting blood samples will be collected for the measurement of CMP, insulin, FFa and two 24-h urine samples will be collected under mineral oil to be analyzed for total volume, pH, Cr, na, K, Ca, Mg, Cl, P, uric acid, nH4+, titratable acidity (Ta), sulfate, HCo3- and citrate. The morning of day 6, patients will undergo dual 123i-BMiPP and 99mTc-MaG3 (99mTc mercaptoacetyltriglycine mertiatide) SPeCT/CT imaging after 12 hrs of fasting. 99mTc-MaG3 (8-10mCi) will be injected intravenously for the flow phase of a standard renal scan which includes dynamic imaging for 2 minutes. an additional 1 minute image will be acquired (the 2-3 minute image on a standard renal scan). acquisition will then stop. immediately afterward 123i-BMiPP (4-5mCi) will be injected intravenously for a 1hour uptake period. after the 1 hour uptake dual isotope (Tc-99m and i-123) SPeCT/CT images of the kidney will be acquired on a clinical Siemens Symbia dual head SPeCT/CT system. The 99mTc-MaG3 flow image data will be used to measure renal plasma flow,12 using the Ge Xeleris renal analysis software package already installed on the clinical SPeCT/CT system. The 123i-BMiPP, a gamma emitter with a half-life of 13.13 hours, is to measure renal 123i-BMiPP (FFa) uptake 13 123i-BMiPP uptake will be corrected for effective renal plasma flow (mL/min) measured with 99mTc-MaG3, using the Ge Xeleris renal analysis software package.

Expected findings: If the hypothesis is correct, the investigators expect increased FFa uptake as measured by 123i-BMiPP SPeCT/CT corrected for renal effective plasma flow in the kidney cortex of iuan patients vs. matched controls.

ELIGIBILITY:
Inclusion Criteria:

* In the IUAN group (N=10), we will include adult subjects with documented IUAN, age > 21 years, either sex, any ethnicity
* In the Control group (N=10), we will include volunteers with no history of stone disease matched for age (within 5 years), gender, ethnicity, BMI (within 10%) and diabetes status

Exclusion Criteria:

* Contraindications to SPECT/CT, pregnancy, breastfeeding, chronic renal disease (eGFR < 60 ml/min/1.73m2), proteinuria, genetic diseases of the kidney, inborn defects of lipid metabolism, alcohol abuse, liver disease (patients with highly elevated total bilirubin, elevated liver enzymes AST, ALT and alkaline phosphatase and those with an established liver disease), anemia, and pharmacological treatment with insulin or insulin-sensitizing drugs such as thiazolidinediones (TZD).
* Patients on antidyslipidemic drugs, alkali therapy or allopurinol will be instructed to discontinue these drugs 2 weeks prior to the study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Increased FFA uptake as measured by 123I-BMIPP SPECT/CT corrected for renal effective plasma flow in the kidney cortex of IUAN patients vs. matched controls | 6 days
  Based on preliminary animal study, we anticipate a mean difference of approximately 26% between IUAN and control non-stone forming subjects, but with a higher CV of 20%. For 80% power (=0.05), will be able to detect at 1.5 standardized effect size (%change/CV) with n=10 per group. Comparisons between IUAN and non-stone former groups will be made with two-sample t-tests or Wilcoxon Rank Sum tests.

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Sakhaee, MD, Principal Investigator — UT Southwestern
Locations (2):
- United States (2):
  - UT Southwestern Medical Center - Center for Mineral Metabolism, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No